CLINICAL TRIAL: NCT04627610
Title: Rate of Recurrence of Dyschezia in Rectal Prolapse, Rectocele and Elytrocele at 10 Years and Over After Rectopexy Intervention.
Brief Title: Recurrence of Dyschezia in Rectal Prolapse, Rectocele and Elytrocele
Acronym: PEXITY
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.290; 2020-A02325-34 (Other: ID RCB)
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rectal prolapse, rectocele and elytrocele — Recurrence of dyschesia on rectal prolapse, rectocele and elytrocele

SUMMARY:
Prolapse of the rectum is a pathology that preferentially affects older women with a significant impact on quality of life. A very large number of therapeutic approaches can be proposed (functional treatment, surgical techniques by perineal approach and surgical techniques by anterior approach).

D'Hoore and Pennix described Ventral Rectopexy with prosthetic reinforcement which is accepted as a standard of treatment in much of Europe for externalized prolapse but remains maligned in much of the world. Due to the relatively recent appearance of this technique and the great variability in the management methods, the long-term results of Ventral Rectopexy have been little studied.

This surgical technique is the preferred approach offered at CHU Grenoble Alpes. Pr Faucheron have internationally recognized experience in surgical grip with a very high patient volume in recent years.

DETAILED DESCRIPTION:
Prolapse of the rectum is a pathology that preferentially affects older women with a significant impact on quality of life. A very large number of therapeutic approaches can be proposed (functional treatment, surgical techniques by perineal approach and surgical techniques by anterior approach).

D'Hoore and Pennix described Ventral Rectopexy with prosthetic reinforcement which is accepted as a standard of treatment in much of Europe for externalized prolapse but remains maligned in much of the world. Due to the relatively recent appearance of this technique and the great variability in the management methods, the long-term results of Ventral Rectopexy have been little studied.

This surgical technique is the preferred approach offered at CHU Grenoble Alpes. Pr Faucheron have internationally recognized experience in surgical grip with a very high patient volume in recent years.

The objective of this work is to describe the long-term results of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated for rectal prolapse or enterocele for 10 or more
* Age 18 and over
* Patients informed

Exclusion Criteria:

- Patient opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patient operated for rectal prolapse or enterocele for 10 or more
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-09-09 (Actual)

PRIMARY OUTCOMES:
rate of recurrence leading to reoperation within 10 years of rectopexy intervention for "rectal prolapse, enterocele or elytrocele". | 10 years
  The rate of re-operations for recurrence of rectal prolapse, enterocele or elytrocele within 10 years of the "index" intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc FAUCHERON, Study Director — CHU Grenoble Alpes; Giorgia Mastronicola, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Hoore A, Cadoni R, Penninckx F. Long-term outcome of laparoscopic ventral rectopexy for total rectal prolapse. Br J Surg. 2004 Nov;91(11):1500-5. doi: 10.1002/bjs.4779. PMID 15499644
- [Background] Faucheron JL, Voirin D, Riboud R, Waroquet PA, Noel J. Laparoscopic anterior rectopexy to the promontory for full-thickness rectal prolapse in 175 consecutive patients: short- and long-term follow-up. Dis Colon Rectum. 2012 Jun;55(6):660-5. doi: 10.1097/DCR.0b013e318251612e. PMID 22595845
- [Background] Faucheron JL, Trilling B, Girard E, Sage PY, Barbois S, Reche F. Anterior rectopexy for full-thickness rectal prolapse: Technical and functional results. World J Gastroenterol. 2015 Apr 28;21(16):5049-55. doi: 10.3748/wjg.v21.i16.5049. PMID 25945021
- [Background] Trilling B, Sage PY, Reche F, Barbois S, Waroquet PA, Faucheron JL. Early experience with ambulatory robotic ventral rectopexy. J Visc Surg. 2018 Feb;155(1):5-9. doi: 10.1016/j.jviscsurg.2017.05.005. Epub 2018 Feb 1. PMID 29396113